CLINICAL TRIAL: NCT02761694
Title: A Phase 1b Study of ARQ 751 as a Single Agent or in Combination With Other Anti-cancer Agents in Adult Subjects With Advanced Solid Tumors With PIK3CA / AKT / PTEN Mutations
Brief Title: Vevorisertib (ARQ 751) as a Single Agent or in Combination With Other Anti-Cancer Agents, in Solid Tumors With PIK3CA / AKT / PTEN Mutations (MK-4440-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4440-001; ARQ 751-101 (Other: ArQule Study Number); MK-4440-001 (Other: Merck)
Record Dates: First submitted 2016-04-29; First posted 2016-05-04 (Estimated); Results first posted 2022-06-15 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Solid Tumors
Keywords: AKT1; AKT2; AKT3; PI3K; solid tumors; cancer; ARQ 751; PTEN
MeSH Terms: conditions — Neoplasms | interventions — Fulvestrant; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- Part 1: Vevorisertib 5 mg QD (Experimental): Participants will receive vevorisertib 5 mg orally once a day (QD) until discontinuation or toxicity.
  Interventions: Drug: Vevorisertib
- Part 1: Vevorisertib 10 mg QD (Experimental): Participants will receive vevorisertib 10 mg orally QD until discontinuation or toxicity.
  Interventions: Drug: Vevorisertib
- Part 1: Vevorisertib 20 mg QD (Experimental): Participants will receive vevorisertib 20 mg orally QD until discontinuation or toxicity.
  Interventions: Drug: Vevorisertib
- Part 1: Vevorisertib 25 mg QD (Experimental): Participants will receive vevorisertib 25 mg orally QD until discontinuation or toxicity.
  Interventions: Drug: Vevorisertib
- Part 1: Vevorisertib 25 mg QOD (Experimental): Participants will receive vevorisertib 25 mg orally every other day (QOD) until discontinuation or toxicity.
  Interventions: Drug: Vevorisertib
- Part 1: Vevorisertib 50 mg QD (Experimental): Participants will receive vevorisertib 50 mg orally QD until discontinuation or toxicity.
  Interventions: Drug: Vevorisertib
- Part 1: Vevorisertib 75 mg QD (Experimental): Participants will receive vevorisertib 75 mg orally QD until discontinuation or toxicity.
  Interventions: Drug: Vevorisertib
- Part 1: Vevorisertib 100 mg QD (Experimental): Participants will receive vevorisertib 100 mg orally QD until discontinuation or toxicity.
  Interventions: Drug: Vevorisertib
- Part 2: Vevorisertib 50 mg QD plus Paclitaxel (Experimental): Participants will receive vevorisertib 50 mg orally QD plus paclitaxel 80 mg/m^2 via intravenous (IV) infusion on Days 1, 7, 15 followed by a week of rest of each 28-day cycle until discontinuation or toxicity.
  Interventions: Drug: Vevorisertib; Drug: Paclitaxel
- Part 2: Vevorisertib 75 mg QD plus Paclitaxel (Experimental): Participants will receive vevorisertib 75 mg orally QD plus paclitaxel 80 mg/m^2 via IV infusion on Days 1, 7, and 15 followed by a week of rest of each 28-day cycle until discontinuation or toxicity.
  Interventions: Drug: Vevorisertib; Drug: Paclitaxel
- Part 2: Vevorisertib 50 mg QD plus Fulvestrant (Experimental): Participants will receive vevorisertib 50 mg orally QD plus fulvestrant 500 mg via intramuscular (IM) injection on Days 1 and 15 of Cycle 1, and Day 1 of each 28-day cycle thereafter until discontinuation or toxicity.
  Interventions: Drug: Vevorisertib; Drug: Fulvestrant
- Part 2: Vevorisertib 75 mg QD plus Fulvestrant (Experimental): Participants will receive vevorisertib 75 mg orally QD plus fulvestrant 500 mg via IM injection on Days 1 and 15 of Cycle 1, and Day 1 of each 28-day cycle thereafter until discontinuation or toxicity.
  Interventions: Drug: Vevorisertib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Vevorisertib — Administered as an oral dose every day or every other day.
  Other Names: ARQ 751; MK-4440
Drug: Fulvestrant — Administered as an intramuscular (IM) injection.
  Other Names: Faslodex
  Arms: Part 2: Vevorisertib 50 mg QD plus Fulvestrant; Part 2: Vevorisertib 75 mg QD plus Fulvestrant
Drug: Paclitaxel — Administered as an intravenous (IV) infusion.
  Other Names: Taxol
  Arms: Part 2: Vevorisertib 50 mg QD plus Paclitaxel; Part 2: Vevorisertib 75 mg QD plus Paclitaxel

SUMMARY:
The primary objectives of this study are: Part 1 - Vevorisertib as single agent: To assess the safety and tolerability of vevorisertib in participants with advanced solid tumors with v-Akt murine thymoma viral oncogene homolog (AKT) 1, 2, 3 genetic alterations, activating phosphatidylinositol-3-kinase (PI3K) mutations, phosphatase and tensin homolog deleted on chromosome ten (PTEN)-null, or other known actionable PTEN mutations; Part 2 - Vevorisertib in combination with other anti-cancer agents: To assess the safety and tolerability of vevorisertib in combination with paclitaxel or fulvestrant in participants with advanced, inoperable, metastatic and/or recurrent solid tumors with phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA) / PTEN actionable mutations and/or AKT genetic alterations.

DETAILED DESCRIPTION:
This study was terminated due to business reasons, and pharmacokinetic (PK) testing was prioritized.

ELIGIBILITY:
Inclusion Criteria

1. Signed written informed consent granted prior to initiation of any study-specific procedures
2. 18 years of age and older
3. Histologically and/or cytologically documented diagnosis of a selected tumor type that is locally advanced, inoperable, metastatic or recurrent (including but not restricted to breast cancer, TNBC [triple negative]; HR-positive [HR+]/HER2-negative [HER2-] or endometrial cancer)
4. Documented AKT genetic alterations or known actionable PIK3CA/PTEN mutations by genetic testing

   • Participants with tumors with PTEN null/PTEN loss-of-function mutations are not eligible
5. For combination arms; participants should be eligible for paclitaxel or fulvestrant therapy as per Investigator assessment
6. Failure to respond to standard systemic therapy, or for whom standard or curative systemic therapy does not exist or is not tolerable

   * Participants in single agent arm (with AKT genetic alterations) and participants in dose escalation cohorts of combination therapy arms should have at least one line of standard systemic therapy
   * Participants in single agent arm (with PIK3CA/PTEN actionable mutations) and participants in the expansion cohorts of combination therapy arms should have no more than 3 prior systemic regimens for the advanced disease
   * Neoadjuvant and adjuvant chemotherapy are considered one regimen if they are a continuation of the same regimen with interval debulking surgery
   * If the participant is refractory or has disease progression within 6 months after completion of the adjuvant treatment, then the adjuvant treatment should be considered as the line of treatment rather than an adjuvant therapy.
   * Endocrine (hormonal) therapy does not count toward total lines of therapy
   * Maintenance therapy is considered part of the preceding regimen if one or more of the same drugs are continued
7. Has at least one measurable target lesion according to RECIST v. 1.1
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1
9. Adequate organ function as indicated by the following laboratory values. (All laboratory tests must be obtained within 14 days prior to the first dose of study treatment):

   1. Hematological

      * Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
      * Platelet count (Plt) ≥ 100 x 10⁹/L
      * Hemoglobin (Hb) ≥ 9 g/dL
      * International normalized ratio (INR) 0.8 to upper limit of normal (ULN) or ≤ 3 for participants receiving anticoagulant therapy such as Coumadin or heparin
   2. Renal

      * Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with serum creatinine levels > 1.5 x institutional ULN
   3. Hepatic

      * Total bilirubin ≤ 1.5 x ULN
      * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN or ≤ 5 x ULN for participants with known liver metastases
   4. Metabolic

      * Glycated hemoglobin (HbA1c) ≤ 8% (≤ 64 mmol/mol)
10. If a participant is currently receiving bisphosphonates or any other drug for treatment of osteoporosis, treatment-induced bone loss and metastases to bone, the participant must have received the bisphosphonates for at least four weeks prior to the first dose of study treatment

    • Initiation of bisphosphonates or similar agents during the study may be allowed provided the participant completes the first cycle of treatment without any dose limiting toxicity (DLT) and the Investigator rules out tumor progression
11. Male or female participants of child-producing potential must agree to use adequate contraception, including double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after the last dose of study treatment
12. Women of childbearing potential must have a negative serum pregnancy test. "Women of childbearing potential" is defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months prior to the first dose of study treatment

Exclusion Criteria

1. Anti-cancer therapy, such as chemotherapy, immunotherapy, hormonal therapy, targeted therapy, or investigational agents within five half-lives or four weeks, whichever is shorter, prior to administration of the first dose of study treatment

   * To be eligible for study treatment, toxicity from prior treatment(s) must recover to Grade ≤ 1, except for alopecia
   * Concurrent systemic high-dose corticosteroids (in dosing exceeding 10 mg QD of prednisone equivalent) when used intermittently in an antiemetic regimen, for central nervous system (CNS) metastases management, or as a part of the premedication regimen are allowed
2. Radiation therapy within four weeks, or palliative radiation therapy within two weeks, prior to administration of the first dose of study treatment

   * To be eligible for study treatment, radiation therapy-related toxicity must recover to Grade ≤ 1 prior to administration of the first dose of study treatment
   * Concurrent palliative radiotherapy for local pain-control or prevention of fracture (for known bone metastases) may be allowed provided the participant completes the first cycle of treatment, does not meet criteria of progressive disease, and treated lesions will not be included in the target/non-target lesion assessment
3. Major surgical procedure within four weeks prior to administration of the first dose of study treatment

   • To be eligible for the study treatment, all surgical wounds must be fully healed, and any surgery-related adverse events must recover to Grade ≤ 1.
4. Unable or unwilling to swallow the complete daily dose of vevorisertib
5. Previous treatment with

   * AKT inhibitors (e.g., ARQ 092, MK-2206, GSK2141795, AZD5363; prior treatment with PI3K or mammalian target of rapamycin (mTOR) inhibitor are allowed)
   * Prior taxane therapy for the advanced, metastatic disease (for participants considered for vevorisertib +paclitaxel combination arm only)
6. Known prior allergic reaction to or severe intolerance of paclitaxel or fulvestrant. Intolerance is defined as a serious adverse event (AE), a grade 3 or 4 AE per Common Terminology Criteria for Adverse Events (CTCAE) v.4.03, or permanent treatment discontinuation
7. History of Type 1 diabetes mellitus or Type 2 diabetes mellitus requiring regular medication (other than oral hypoglycemic agents) or fasting glucose ≥ 160 mg/dL at Screening visit
8. Significant gastrointestinal disorder(s) that could, in the opinion of the Investigator, interfere with the absorption, metabolism, or excretion of vevorisertib (e.g., inflammatory bowel disease, Crohn's disease, ulcerative colitis, extensive gastric resection)
9. Known untreated or active CNS metastases and/or carcinomatous meningitis

   • To be eligible for the study treatment, participants must have stable disease ≥ 1 month, confirmed by magnetic resonance imaging (MRI) or computed tomography (CT) scan, and have CNS metastases well controlled by low-dose steroids, anti-epileptics, or other symptom-relieving medications
10. History of myocardial infarction (MI) or New York Heart Association (NYHA) Class II-IV congestive heart failure within 6 months of the administration of the first dose of study treatment (MI occurring > 6 months of the first dose of study treatment will be permitted); Grade 2 or worse conduction defect (e.g., right or left bundle branch block)
11. A heart rate corrected QT (QTc) interval ≥ 480 msec, using the Fridericia's formula QTcF
12. Left ventricular ejection fraction (LVEF) <50% as determined by Multiple Gated Acquisition (MUGA) scan or echocardiogram (ECHO) in participants who received prior treatment with anthracyclines
13. Concurrent severe and/or uncontrolled illness not related to cancer and/or social situation that would limit compliance with study requirements, including but not limited to:

    * Psychiatric illness, substance abuse
    * Ongoing or active known infection, including human immunodeficiency virus (HIV) infection, hepatitis B or C virus
    * Significant pulmonary dysfunction, including pneumonitis, interstitial lung disease (ILD), idiopathic pulmonary fibrosis, cystic fibrosis, severe chronic obstructive pulmonary disease (COPD)
    * Peripheral neuropathy grade ≥2 (vevorisertib+paclitaxel combination arm)
    * Bleeding diathesis, thrombocytopenia or coagulation disorders (vevorisertib+fulvestrant combination arm)
    * Thrombotic/coagulation disorders within 6 months prior to the first dose of study treatment unless stable on anticoagulation for > 3 months
14. Active or history of other malignancy other than the current cancer within 2 years of the first dose of study treatment, with the exception of carcinoma in-situ of the cervix, basal cell carcinoma, and superficial bladder tumors curatively treated
15. Blood transfusion or administration of growth factors within 5 days prior to a blood draw being used to confirm eligibility
16. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-06-26 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (6):
- United States (6):
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Charleston Hematology Oncology, Charleston, South Carolina
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Pant S, Hamilton E, Ulahannan SV, Strauss JF, Braiteh FS, Huang M, Liaw DCH. Phase 1b study of pan-AKT inhibitor vevorisertib alone or with paclitaxel or fulvestrant in PIK3CA/AKT/PTEN-mutated advanced solid tumors. Cancer. 2023 Jun 15;129(12):1919-1929. doi: 10.1002/cncr.34733. Epub 2023 Mar 27. PMID 36970876

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Vevorisertib 5 mg QD: Participants received vevorisertib 5 mg orally once a day (QD) until discontinuation or toxicity.
- Part 1: Vevorisertib 10 mg QD: Participants received vevorisertib 10 mg orally QD until discontinuation or toxicity.
- Part 1: Vevorisertib 20 mg QD: Participants received vevorisertib 20 mg orally QD until discontinuation or toxicity.
- Part 1: Vevorisertib 25 mg QD: Participants received vevorisertib 25 mg orally QD until discontinuation or toxicity.
- Part 1: Vevorisertib 25 mg QOD: Participants received vevorisertib 25 mg orally every other day (QOD) until discontinuation or toxicity.
- Part 1: Vevorisertib 50 mg QD: Participants received vevorisertib 50 mg orally QD until discontinuation or toxicity.
- Part 1: Vevorisertib 75 mg QD: Participants received vevorisertib 75 mg orally QD until discontinuation or toxicity.
- Part 1: Vevorisertib 100 mg QD: Participants received vevorisertib 100 mg orally QD until discontinuation or toxicity.
- Part 2: Vevorisertib 50 mg QD Plus Paclitaxel: Participants received vevorisertib 50 mg orally QD plus paclitaxel 80 mg/m^2 via intravenous (IV) infusion on Days 1, 7, 15 followed by a week of rest of each 28-day cycle until discontinuation or toxicity.
- Part 2: Vevorisertib 75 mg QD Plus Paclitaxel: Participants received vevorisertib 75 mg orally QD plus paclitaxel 80 mg/m^2 via IV infusion on Days 1, 7, and 15 followed by a week of rest of each 28-day cycle until discontinuation or toxicity.
- Part 2: Vevorisertib 50 mg QD Plus Fulvestrant: Participants received vevorisertib 50 mg orally QD plus fulvestrant 500 mg via intramuscular (IM) injection on Days 1 and 15 of Cycle 1, and Day 1 of each 28-day cycle thereafter until discontinuation or toxicity.
- Part 2: Vevorisertib 75 mg QD Plus Fulvestrant: Participants received vevorisertib 75 mg orally QD plus fulvestrant 500 mg via IM injection on Days 1 and 15 of Cycle 1, and Day 1 of each 28-day cycle thereafter until discontinuation or toxicity.
Period: Overall Study
Arm/Group | Part 1: Vevorisertib 5 mg QD | Part 1: Vevorisertib 10 mg QD | Part 1: Vevorisertib 20 mg QD | Part 1: Vevorisertib 25 mg QD | Part 1: Vevorisertib 25 mg QOD | Part 1: Vevorisertib 50 mg QD | Part 1: Vevorisertib 75 mg QD | Part 1: Vevorisertib 100 mg QD | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant
Started | 4 | 4 | 1 | 3 | 3 | 3 | 33 | 8 | 5 | 5 | 3 | 6
Treated | 4 | 4 | 1 | 3 | 3 | 3 | 32 | 8 | 5 | 5 | 3 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 1 | 3 | 3 | 3 | 33 | 8 | 5 | 5 | 3 | 6
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 1 | 1 | 4
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Other | 4 | 4 | 1 | 2 | 3 | 3 | 18 | 8 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Vevorisertib 5 mg QD | Part 1: Vevorisertib 10 mg QD | Part 1: Vevorisertib 20 mg QD | Part 1: Vevorisertib 25 mg QD | Part 1: Vevorisertib 25 mg QOD | Part 1: Vevorisertib 50 mg QD | Part 1: Vevorisertib 75 mg QD | Part 1: Vevorisertib 100 mg QD | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant | Total
Number analyzed (Participants) | 4 | 4 | 1 | 3 | 3 | 3 | 33 | 8 | 5 | 5 | 3 | 6 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (11.5) | 57.0 (14.4) | 65.0 (NA) — Standard deviation was not calculatable when n<2. | 62.0 (3.6) | 58.3 (11.6) | 53.0 (20.2) | 58.6 (11.9) | 59.0 (8.4) | 57.2 (19.7) | 59.8 (11.3) | 52.3 (7.6) | 65.8 (5.6) | 59.0 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 0 | 3 | 3 | 3 | 19 | 7 | 5 | 2 | 3 | 6 | 56
  Male | 1 | 2 | 1 | 0 | 0 | 0 | 14 | 1 | 0 | 3 | 0 | 0 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 3 | 4 | 1 | 3 | 3 | 3 | 31 | 7 | 5 | 5 | 3 | 6 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 6
  White | 4 | 3 | 1 | 3 | 3 | 3 | 30 | 6 | 5 | 4 | 3 | 6 | 71
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with study-drug treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to approximately 120 weeks
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Vevorisertib 20 mg: Participants received vevorisertib 20 mg orally QD until discontinuation or toxicity.
Arm/Group | Part 1: Vevorisertib 5 mg QD | Part 1: Vevorisertib 10 mg QD | Part 1: Vevorisertib 20 mg | Part 1: Vevorisertib 25 mg QD | Part 1: Vevorisertib 25 mg QOD | Part 1: Vevorisertib 50 mg QD | Part 1: Vevorisertib 75 mg QD | Part 1: Vevorisertib 100 mg QD | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant
Number analyzed (Participants) | 4 | 4 | 1 | 3 | 3 | 3 | 32 | 8 | 5 | 5 | 3 | 6
Participants | 4 | 4 | 1 | 3 | 3 | 3 | 32 | 8 | 5 | 5 | 3 | 6

2. Primary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: as for outcome 1
Time Frame: Up to approximately 116 weeks
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Vevorisertib 5 mg QD | Part 1: Vevorisertib 10 mg QD | Part 1: Vevorisertib 20 mg QD | Part 1: Vevorisertib 25 mg QD | Part 1: Vevorisertib 25 mg QOD | Part 1: Vevorisertib 50 mg QD | Part 1: Vevorisertib 75 mg QD | Part 1: Vevorisertib 100 mg QD | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant
Number analyzed (Participants) | 4 | 4 | 1 | 3 | 3 | 3 | 32 | 8 | 5 | 5 | 3 | 6
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 1

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Vevorisertib
Description: Cmax was defined as the maximum plasma drug concentration. This study was terminated because of business reasons. Due to study termination, pharmacokinetic (PK) testing was prioritized for dosing arms and timepoints that would provide the required data to support programmatic decision-making and subsequent clinical studies. Zero participants analyzed entered in the table indicate data were not generated and no data were available. Cmax is reported as geometric mean with a percent coefficient of variation.
Time Frame: Cycle 1 Day 1: predose and 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose; Cycle 1 Day 22: predose and 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose; Cycle 2 Day 1: predose. Cycle = 28 days.
Population: All participants who received at least 1 dose of study drug and had ≥1 sample collected to assess Cmax at each time point. Due to termination of the study, PK testing was prioritized for dosing arms and time points that would support programmatic decision-making and subsequent clinical studies. Zero participants analyzed indicate data were not generated and no data were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Vevorisertib 5 mg QD | Part 1: Vevorisertib 10 mg QD | Part 1: Vevorisertib 20 mg QD | Part 1: Vevorisertib 25 mg QD | Part 1: Vevorisertib 25 mg QOD | Part 1: Vevorisertib 50 mg QD | Part 1: Vevorisertib 75 mg QD | Part 1: Vevorisertib 100 mg QD | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant
Number analyzed (Participants) | 2 | 3 | 1 | 3 | 3 | 3 | 28 | 8 | 4 | 4 | 3 | 6
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 2 | 1 | 3 | 2 | 3 | 28 | 8 | 3 | 4 | 1 | 6
  Cycle 1 Day 1 | NA (NA) — Geometric Mean (percent geometric coefficient of variation) were not calculable because levels were below the limit of quantification (BLQ). | 4.820 (80.1) | 15.3 (NA) — Percent Geometric Coefficient of Variation was not calculable when n<2. | 51.39 (68.1) | 22.73 (5.9) | 59.79 (7.6) | 98.75 (88.2) | 122.6 (107.1) | 29.13 (245.6) | 49.11 (67.0) | 91.7 (NA) — Percent Geometric Coefficient of Variation was not calculable when n<2. | 166.7 (101.7)
  Cycle 1 Day 22: number analyzed (Participants) | 2 | 3 | 1 | 3 | 3 | 3 | 11 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Day 22 | 4.154 (45.3) | 12.82 (71.1) | 7.79 (NA) — Percent Geometric Coefficient of Variation was not calculable when n<2. | 65.40 (61.5) | 19.49 (96.5) | 55.15 (76.7) | 225.1 (80.0) | 207.7 (80.6) |  |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 4 | 2 | 3 | 5
  Cycle 2 Day 1 |  |  |  |  |  |  | 186.8 (47.3) |  | 78.36 (216.8) | 79.52 (69.6) | 62.59 (140.1) | 138.2 (48.4)

4. Secondary Outcome: Area Under the Curve From 0-24 Hours (AUC0-24 Hours) of Vevorisertib
Description: AUC0-24hrs was defined as area under the concentration-time curve from time 0 to 24 hours after dose administration. This study was terminated because of business reasons. Due to study termination, pharmacokinetic (PK) testing was prioritized for dosing arms and timepoints that would provide the required data to support programmatic decision-making and subsequent clinical studies. Zero participants analyzed entered in the table indicate data were not generated and no data were available. AUC0-24 is reported as geometric mean with a percent coefficient of variation.
Time Frame: as for outcome 3
Population: All participants who received at least 1 dose of study drug and had ≥1 sample collected to assess AUC0-24 at each time point. Due to termination of the study, PK testing was prioritized for dosing arms and time points that would support programmatic decision-making and subsequent clinical studies. Zero participants analyzed indicate data were not generated and no data were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Part 1: Vevorisertib 5 mg QD | Part 1: Vevorisertib 10 mg QD | Part 1: Vevorisertib 20 mg QD | Part 1: Vevorisertib 25 mg QD | Part 1: Vevorisertib 25 mg QOD | Part 1: Vevorisertib 50 mg QD | Part 1: Vevorisertib 75 mg QD | Part 1: Vevorisertib 100 mg QD | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant
Number analyzed (Participants) | 2 | 2 | 1 | 3 | 3 | 3 | 28 | 8 | 4 | 3 | 3 | 6
hours*ng/mL
  Cycle 1 Day1: number analyzed (Participants) | 2 | 1 | 1 | 3 | 2 | 3 | 28 | 8 | 1 | 3 | 1 | 6
  Cycle 1 Day1 | NA (NA) — Geometric Mean (percent geometric coefficient of variation) were not calculable because levels were below the limit of quantification (BLQ). | 12.27 (NA) — Percent Geometric Coefficient of Variation was not calculable when n<2. | 42.2 (NA) — Percent Geometric Coefficient of Variation was not calculable when n<2. | 244.1 (113.3) | 128.6 (52.4) | 287.5 (4.5) | 667.6 (84.6) | 786.1 (117.7) | 391.1 (NA) — Percent Geometric Coefficient of Variation was not calculable when n<2. | 649.6 (41.7) | 449 (NA) — Percent Geometric Coefficient of Variation was not calculable when n<2. | 1115 (73.5)
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 2 | 1 | 3 | 3 | 3 | 11 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Day 22 |  | 67.89 (197.1) | 78.5 (NA) — Percent Geometric Coefficient of Variation was not calculable when n<2. | 501.8 (35.5) | 181.2 (59.0) | 543.8 (78.2) | 1832 (68.5) | 1786 (82.4) |  |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 4 | 2 | 3 | 3
  Cycle 2 Day 1 |  |  |  |  |  |  | 2013 (66.4) |  | 837.2 (200.6) | 1280 (39.1) | 750.7 (67.0) | 1948 (49.7)

5. Secondary Outcome: Elimination Half-life (t½) of Vevorisertib
Description: t1/2 was defined as the terminal elimination half-life of drug. This study was terminated because of business reasons. Due to study termination, pharmacokinetic (PK) testing was prioritized for dosing arms and timepoints that would provide the required data to support programmatic decision-making and subsequent clinical studies. Zero participants analyzed entered in the table indicate data were not generated and no data were available. t1/2 is reported as geometric mean with a percent coefficient of variation.
Time Frame: Cycle 1 Day 1: predose, 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose; Cycle 1 Day 22: predose, 1, 2, 4, 6, 8, 10, 12, and 24 hours postdose; Cycle 2 Day 1: predose. Cycle = 28 days.
Population: All participants who received at least 1 dose of study drug and had ≥1 sample collected to assess t1/2 at each time point. Due to termination of the study, PK testing was prioritized for dosing arms and time points that would support programmatic decision-making and subsequent clinical studies. Zero participants analyzed indicate data were not generated and no data were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1: Vevorisertib 5 mg QD | Part 1: Vevorisertib 10 mg QD | Part 1: Vevorisertib 20 mg QD | Part 1: Vevorisertib 25 mg QD | Part 1: Vevorisertib 25 mg QOD | Part 1: Vevorisertib 50 mg QD | Part 1: Vevorisertib 75 mg QD | Part 1: Vevorisertib 100 mg QD | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant
Number analyzed (Participants) | 2 | 2 | 1 | 3 | 2 | 3 | 25 | 7 | 3 | 3 | 2 | 6
hours
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 0 | 1 | 3 | 2 | 3 | 25 | 7 | 1 | 3 | 1 | 6
  Cycle 1 Day 1 | NA (NA) — Geometric Mean (percent geometric coefficient of variation) were not calculable because levels were below the limit of quantification (BLQ). |  | 3.68 (NA) — Percent Geometric Coefficient of Variation was not calculable when n<2. | 15.43 (104.2) | 8.257 (102.7) | 15.94 (19.3) | 12.39 (37.7) | 7.437 (69.0) | 8.920 (NA) — Percent Geometric Coefficient of Variation was not calculable when n<2. | 8.909 (16.3) | 9.48 (NA) — Percent Geometric Coefficient of Variation was not calculable when n<2. | 9.176 (46.7)
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 2 | 0 | 3 | 2 | 2 | 9 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Day 22 |  | 10.12 (87.0) |  | 39.33 (48.6) | 21.25 (13.8) | 20.03 (1.6) | 12.94 (71.8) | 24.59 (6.9) |  |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 0 | 2 | 1
  Cycle 2 Day 1 |  |  |  |  |  |  | 22.93 (36.8) |  | 20.89 (70.9) |  | 28.78 (16.3) | 11.46 (NA) — Percent Geometric Coefficient of Variation was not calculable when n<2.

6. Secondary Outcome: Number of Participants With a Dose-Limiting Toxicity (DLT), for the Determination of Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D)
Description: DLTs consisted of hematologic or non-hematologic toxicities. Hematologic DLT was any grade (Gr) 4 anemia, Gr 4 neutropenia, Gr 4 thrombocytopenia, Gr 3 lasting >7 days, Gr 3 thrombocytopenia in the presence of bleeding, or ≥ Gr 3 hyperglycemia. Non-hematologic DLT was any Gr 3, 4 or 5 non-hematologic toxicity with the exception of: (1) Gr 3 nausea, vomiting, diarrhea or responding to optimal medical management within 48 hours; (2) alopecia. Per protocol DLTs were analyzed in the first 28-day treatment cycle. The number of participants experiencing DLTs is reported here for all participants who got ≥1 dose of study drug.
Time Frame: Cycle 1 (Up to approximately 28 days)
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Vevorisertib 5 mg QD | Part 1: Vevorisertib 10 mg QD | Part 1: Vevorisertib 20 mg QD | Part 1: Vevorisertib 25 mg QD | Part 1: Vevorisertib 25 mg QOD | Part 1: Vevorisertib 50 mg QD | Part 1: Vevorisertib 75 mg QD | Part 1: Vevorisertib 100 mg QD | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant
Number analyzed (Participants) | 4 | 4 | 1 | 3 | 3 | 3 | 32 | 8 | 5 | 5 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0

7. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who have best response of Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
Time Frame: Up to approximately 116 weeks
Population: All participants who received at least 1 dose of study treatment and had ORR data available.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1: Vevorisertib 5 mg QD | Part 1: Vevorisertib 10 mg QD | Part 1: Vevorisertib 20 mg QD | Part 1: Vevorisertib 25 mg QD | Part 1: Vevorisertib 25 mg QOD | Part 1: Vevorisertib 50 mg QD | Part 1: Vevorisertib 75 mg QD | Part 1: Vevorisertib 100 mg QD | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant
Number analyzed (Participants) | 3 | 3 | 1 | 3 | 3 | 2 | 24 | 7 | 4 | 3 | 2 | 4
Percentage of Participants | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 0 [0.00 to 97.50] | 33.3 [0.84 to 90.57] | 0 [0.00 to 70.76] | 0 [0.00 to 84.19] | 4.2 [0.11 to 21.12] | 14.3 [0.36 to 57.87] | 50.0 [6.76 to 93.24] | 0 [0.00 to 70.76] | 0 [0.00 to 84.19] | 0 [0.00 to 60.24]

8. Secondary Outcome: Best Overall Response (BOR)
Description: BOR was assessed using RECIST 1.1. Response categories included: CR: disappearance of all target lesions; PR: at least a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD; Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; and Inevaluable: participants who have SD as their best overall response but fail to achieve the protocol-defined duration for SD. Percentage of participants with CR, PR, SD, PD, or inevaluable as a best overall response have been reported.
Time Frame: Up to approximately 116 weeks
Population: All participants who received at least 1 dose of study treatment and had BOR data available.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1: Vevorisertib 5 mg QD | Part 1: Vevorisertib 10 mg QD | Part 1: Vevorisertib 20 mg QD | Part 1: Vevorisertib 25 mg QD | Part 1: Vevorisertib 25 mg QOD | Part 1: Vevorisertib 50 mg QD | Part 1: Vevorisertib 75 mg QD | Part 1: Vevorisertib 100 mg QD | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant
Number analyzed (Participants) | 3 | 3 | 1 | 3 | 3 | 2 | 24 | 7 | 4 | 3 | 2 | 4
Percentage of Participants
  Complete Response (CR) | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 0 [0.00 to 97.50] | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 0 [0.00 to 84.19] | 0 [0.00 to 14.25] | 0 [0.00 to 40.96] | 0 [0.00 to 60.24] | 0 [0.00 to 70.76] | 0 [0.00 to 84.19] | 0 [0.00 to 60.24]
  Partial Response (PR) | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 0 [0.00 to 97.50] | 33.3 [0.84 to 90.57] | 0 [0.00 to 70.76] | 0 [0.00 to 84.19] | 4.2 [0.11 to 21.12] | 14.3 [0.36 to 57.87] | 50.0 [6.76 to 93.24] | 0 [0.00 to 70.76] | 0 [0.00 to 84.19] | 0 [0.00 to 60.24]
  Stable Disease (SD) | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 100.0 [2.50 to 100.00] | 66.7 [9.43 to 99.16] | 33.3 [0.84 to 90.57] | 50.0 [1.26 to 98.74] | 41.7 [22.11 to 63.36] | 42.9 [9.90 to 81.59] | 25.0 [0.63 to 80.59] | 33.3 [0.84 to 90.57] | 0 [0.00 to 84.19] | 50.0 [6.76 to 93.24]
  Progressive Disease (PD) | 100.0 [29.24 to 100.00] | 100.0 [29.24 to 100.00] | 0 [0.00 to 97.50] | 0 [0.00 to 70.76] | 66.7 [9.43 to 99.16] | 50.0 [1.26 to 98.74] | 54.2 [32.82 to 74.45] | 28.6 [3.67 to 70.96] | 0 [0.00 to 60.24] | 66.7 [9.43 to 99.16] | 100.0 [15.81 to 100.00] | 50.0 [6.76 to 93.24]
  Inevaluable | 0 [0.00 to 70.76] | 0 [0.00 to 0.76] | 0 [0.00 to 97.50] | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 0 [0.00 to 84.19] | 0 [0.00 to 14.25] | 14.3 [0.36 to 57.87] | 25.0 [0.63 to 80.59] | 0 [0.00 to 70.76] | 0 [0.00 to 84.19] | 0 [0.00 to 60.24]

9. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined, per RECIST 1.1, as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) or Stable Disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD].
Time Frame: Up to approximately 116 weeks
Population: All participants who received at least 1 dose of study treatment and had DCR data available.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1: Vevorisertib 5 mg QD | Part 1: Vevorisertib 10 mg QD | Part 1: Vevorisertib 20 mg QD | Part 1: Vevorisertib 25 mg QD | Part 1: Vevorisertib 25 mg QOD | Part 1: Vevorisertib 50 mg QD | Part 1: Vevorisertib 75 mg QD | Part 1: Vevorisertib 100 mg QD | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant
Number analyzed (Participants) | 3 | 3 | 1 | 3 | 3 | 2 | 24 | 7 | 4 | 3 | 2 | 4
Percentage of Participants | 0 [0.00 to 70.76] | 0 [0.00 to 70.76] | 100.0 [2.50 to 100.00] | 100.0 [29.24 to 100.00] | 33.3 [0.84 to 90.57] | 50.0 [1.26 to 98.74] | 45.8 [25.55 to 67.18] | 57.1 [18.41 to 90.10] | 75.0 [19.41 to 99.37] | 33.3 [0.84 to 90.57] | 0 [0.00 to 84.19] | 50.0 [6.76 to 93.24]

ADVERSE EVENTS:
Time Frame: Up to approximately 120 weeks
Description: The analysis population for All-Cause Mortality included all randomized participants.The analysis population for AEs included all randomized participants who received at least 1 dose of study treatment.
Arm/Group | Part 1: Vevorisertib 5 mg QD | Part 1: Vevorisertib 10 mg QD | Part 1: Vevorisertib 20 mg QD | Part 1: Vevorisertib 25 mg QD | Part 1: Vevorisertib 25 mg QOD | Part 1: Vevorisertib 50 mg QD | Part 1: Vevorisertib 75 mg QD | Part 1: Vevorisertib 100 mg QD | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant
All-Cause Mortality (participants affected / at risk) | 2/4 | 2/4 | 0/1 | 1/3 | 0/3 | 1/3 | 7/33 | 2/8 | 2/5 | 2/5 | 1/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/4 | 0/1 | 2/3 | 1/3 | 2/3 | 12/32 | 5/8 | 3/5 | 2/5 | 0/3 | 3/6
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 1/1 | 3/3 | 3/3 | 3/3 | 32/32 | 8/8 | 5/5 | 5/5 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Vevorisertib 5 mg QD (N=4) | Part 1: Vevorisertib 10 mg QD (N=4) | Part 1: Vevorisertib 20 mg QD (N=1) | Part 1: Vevorisertib 25 mg QD (N=3) | Part 1: Vevorisertib 25 mg QOD (N=3) | Part 1: Vevorisertib 50 mg QD (N=3) | Part 1: Vevorisertib 75 mg QD (N=32) | Part 1: Vevorisertib 100 mg QD (N=8) | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel (N=5) | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel (N=5) | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant (N=3) | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Vevorisertib 5 mg QD (N=4) | Part 1: Vevorisertib 10 mg QD (N=4) | Part 1: Vevorisertib 20 mg QD (N=1) | Part 1: Vevorisertib 25 mg QD (N=3) | Part 1: Vevorisertib 25 mg QOD (N=3) | Part 1: Vevorisertib 50 mg QD (N=3) | Part 1: Vevorisertib 75 mg QD (N=32) | Part 1: Vevorisertib 100 mg QD (N=8) | Part 2: Vevorisertib 50 mg QD Plus Paclitaxel (N=5) | Part 2: Vevorisertib 75 mg QD Plus Paclitaxel (N=5) | Part 2: Vevorisertib 50 mg QD Plus Fulvestrant (N=3) | Part 2: Vevorisertib 75 mg QD Plus Fulvestrant (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (5) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Refraction disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 2 (6) | 1 (2) | 2 (3) | 19 (44) | 6 (12) | 1 (6) | 2 (3) | 3 (5) | 2 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (6) | 1 (1) | 2 (5) | 1 (1) | 1 (1) | 8 (13) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (4)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 9 (12) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 3 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 3 (3) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 8 (8) | 2 (3) | 1 (2) | 2 (7) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (7) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 3 (3)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (5) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 10 (11) | 3 (4) | 2 (3) | 1 (1) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Early satiety (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (8) | 2 (2) | 2 (3) | 2 (3) | 1 (1) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cranial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tone disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reflexes abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 5 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (17) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (13) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator agrees not to independently publish the findings except as part of an overall multi-center publication, unless specifically approved in writing by the Sponsor or unless more than 12 months have elapsed since the last participant in the study has completed study treatment.

DOCUMENTS (2):
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT02761694/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT02761694/SAP_001.pdf